CLINICAL TRIAL: NCT07366970
Title: Is There a Benefit From Addition of Exercise in Diabetic Patients With ED Who Complain Low Vitamin D?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB000-14233-64
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus; Erectile Dysfunction; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus; Erectile Dysfunction; Vitamin D Deficiency | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): twenty diabetic men (type 2) who complain presence of low vitamin D and impotence will be pharmacologically treated by administration of Cholecalciferol 200.000 I.U (will be taken every two weeks). this treatment will last for 12 weeks. Additionally, Group number I will perform treadmill walking (one hour walking) with moderate intensity. This walking will be performed three times per designed week for twelve weeks.
  Interventions: Behavioral: exercise and vitamin D intake
- group number 2 (Active Comparator): twenty diabetic men (type 2) who complain presence of low vitamin D and impotence will be pharmacologically treated by administration of Cholecalciferol 200.000 I.U (will be taken every two weeks). this treatment will last for 12 weeks.
  Interventions: Other: vitamin D intake

INTERVENTIONS:
Behavioral: exercise and vitamin D intake — twenty diabetic men (type 2) who complain presence of low vitamin D and impotence will be pharmacologically treated by administration of Cholecalciferol 200.000 I.U (will be taken every two weeks). this treatment will last for 12 weeks. Additionally, Group number I will perform treadmill walking (one hour walking) with moderate intensity. This walking will be performed three times per designed week for twelve weeks.
  Arms: group number 1
Other: vitamin D intake — twenty diabetic men (type 2) who complain presence of low vitamin D and impotence will be pharmacologically treated by administration of Cholecalciferol 200.000 I.U (will be taken every two weeks). this treatment will last for 12 weeks.
  Arms: group number 2

SUMMARY:
males with diabetes complain impotence in the presence of low vitamin D deficiency. pharacmological treatment of low vitamin D levels is necessary but changing lifestyle by performing exercise is also important

DETAILED DESCRIPTION:
forty diabetic men (type 2) who complain presence of low vitamin D and impotence will be divided to group number I and group number II. Both groups will be pharmacologically treated by administration of Cholecalciferol 200.000 I.U (will be taken every two weeks). this treatment will last for 12 weeks. Additionally, Group number I will perform treadmill walking (one hour walking) with moderate intensity. This walking will be performed three times per designed week for twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* diabetic men (forty)
* type 2 diabetes
* complaint of erectile dysfucntion (chronic complaint more than 24 months)
* men with low vitamin D (deiciency in vitamin D)

Exclusion Criteria:

* cardiac patients
* respiratory disease patients
* renal disease
* liver disease

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
international index of erectile function | it will be measured after 12 weeks
  questionnaire used to assess impotence

SECONDARY OUTCOMES:
glycated hemoglubin | It will be measured after 12 weeks
  it will be used to assess blood glcuose
fasting blood glcuose | It will be measured after 12 weeks
  it will be used to assess blood glcuose in serum
body mass index | It will be measured after 12 weeks
  it will be measured on empty stomach and bladder
wasit circumference | it will be measured after 12 weeks
  it will be measured at umbilicus level
high density lipoprotein | It will be measured after 12 weeks
  it will be measured in serum
low density lipoprotein | It will be measured after 12 weeks
  it will be measured in serum
triglycerides | It will be measured after 12 weeks
  it will be assessed in serum
cholesterol | It will be measured after 12 weeks
  it will be assessed in serum
25-hydroxyvitamin D | It will be measured after 12 weeks
  it will be assessed in serum as a metabolite of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Dokki, Giza Governorate, Egypt